CLINICAL TRIAL: NCT03297073
Title: Paracetamol Metabolism Research in Postoperative Hepatic Surgery
Acronym: PARAFOI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015_61; 2016-002632-32 (Other: ID-RCB number)
Record Dates: First submitted 2017-09-25; First posted 2017-09-29 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2021-03

CONDITIONS: Paracetamol Causing Adverse Effects in Therapeutic Use; Hepatic Disease
MeSH Terms: conditions — Digestive System Diseases | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- major hepatic surgery (Experimental): resection greater than or equal to three hepatic segments
  Interventions: Drug: paracetamol; Procedure: hepatic surgery
- hepatic surgery (Experimental): resection less than three hepatic segments
  Interventions: Drug: paracetamol; Procedure: hepatic surgery
- hepatic surgery recovery (Experimental)
  Interventions: Drug: paracetamol; Procedure: hepatic surgery

INTERVENTIONS:
Drug: paracetamol — Paracetamol 1000 mg will be administered 30 minutes before the end of the procedure and then every 6 hours systematically at the following times: 6h / 12h / 18h / 00h.
  The analgesic treatment after hepatectomy with paracetamol will be maintained for at least 5 days in all patients in parenteral form
Procedure: hepatic surgery

SUMMARY:
The main objective of this study was to evaluate the 5-day kinetics of plasma paracetamol levels in postoperative major hepatic surgery (resection greater than or equal to three hepatic segments) compared with less extensive liver resection and hepatic re-intervention. The clearance of indocyanine green is a marker of hepatic perfusion but also of the proper hepatocyte functioning, if hemodynamic conditions are stable.

Some patients may be operated on up to four or five times in the liver. Moreover, these patients probably present an increased risk of postoperative hepatocellular insufficiency due to a quantitative and qualitative decrease in their hepatic parenchyma. It is therefore interesting to evaluate the use of paracetamol in this situation.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring surgery for hepatic resection by initiation under chest or laparoscopic without hepatocellular insufficiency,
* ASA score 1 to 3 (American Society of Anesthesiologists score ranging from 1 to 5 evaluating the preoperative health status of a patient),
* Verification of the understanding of the protocol,

Exclusion Criteria:

* Patients classified ASA 4 or 5,
* Allergy or intolerance to indocyanine green
* Allergy or intolerance to paracetamol,
* Taking of paracetamol the week before the intervention,
* Patient less than 60 Kgs (because decrease of doses of paracetamol),
* Emergency surgery, palliative surgery and surgical recovery,
* Psychic disorder,
* Contra-indication to a treatment used during the study,
* incapable major,
* Intellectual incapacity preventing proper understanding of the protocol,
* Pregnant or nursing woman,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-11-20 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Dosing and kinetics of paracetamolemia | during the 5 post-operative days
  this determination of the plasma paracetamol dosage on D0 (H6: 6 hours after the end of the procedure) and D1 D2 D3 D4 D5 (samples taken at 6 am each day just before the injection of paracetamol whose administration hours will be 6h 12h 18h and midnight)

SECONDARY OUTCOMES:
Dosage of urinary metabolites of paracetamol (paracetamol sulphate, paracetamol glucuronide) | At Day 1, day 3, day 5 post operative
Dosage of N-acetyl-cysteinyl paracetamol ( NAPQI) | At Day 1, day 3, day 5 post operative
Percentage of patients with paracetamolemia greater than 60 mg / mL | during the 5 post-operative days
  60mj/ml = paracetamol toxicity threshold according to Prescott diagram to 6 hours
Plasma Disappearance Rate of indocyanine green (TDP-ICG) by LiMon® | At Day 1, day 3, day 5 post operative
Rate of postoperative hepatocellular insufficiency | at day 5
  The postoperative hepatocellular insufficiency according to the 50/50 criteria (TP <50% and bilirubinemia> 50 μmol / L on the 5th day) according to the type of hepatic resection (with or without clamping, continuous or discontinuous, duration intervention).
Occurrence of complications related to hepatic failure | at day 5
  the complications related to hepatic failure not falling within the "50/50" criteria: jaundice, hepatic encephalopathy, coagulation disorders, ascites, cytolysis, cholestasis.
  Other medical and surgical. Duration of hospitalization in perioperative intensive care and duration of total hospitalization.
  Mortality at 30 days.
Duration of hospitalization in perioperative intensive care | at 30 days
Duration of total hospitalization. | at 30 days
Mortality | at 30 days
Composite characteristics of surgery. | at 30 days
  Characteristics of surgery: duration of intervention, numbers, duration and types of vascular clamping, detailed description of the type of liver resection performed, quantification of bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Lebuffe, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Huriez, CHRU, Lille, France

IPD SHARING:
Plan to Share IPD: No